CLINICAL TRIAL: NCT04074369
Title: Evaluation of CRISPR-based Test for the Rapid Identification of Mycobacterium Tuberculosis Complex in Pulmonary Tuberculosis Suspects
Brief Title: Evaluation of CRISPR-based Test for the Rapid Identification of TB in Pulmonary Tuberculosis Suspects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Wenzhou Central Hospital (Other); Red Cross Hospital, Hangzhou, China (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: 20190601
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Tuberculosis Suspects: Individuals with suspected TB infection
  Interventions: Diagnostic Test: CRISPR-based Test

INTERVENTIONS:
Diagnostic Test: CRISPR-based Test — CRISPR-based Test performed on sputum or BALF in TB suspects.

SUMMARY:
This observational Mycobacterium tuberculosis (MTB) diagnostics evaluation study is a prospective study of pulmonary TB suspects who are undergoing sputum or bronchoalveolar lavage fluid (BALF) evaluation for pulmonary TB. The sensitivity and specificity of the CRISPR-based assay will be compared to clinical diagnosis, conventional culture methods and Xpert MTB/RIF assay on same batch specimens.

ELIGIBILITY:
Inclusion Criteria:

* Suspected pulmonary TB.
* Ability and willingness of candidate or legal guardian/representative to provide informed consent.
* Men and women age equal to or greater than 18 years.

Exclusion Criteria:

* Either receipt of ≥48 cumulative hours OR three or more doses of anti-TB treatment within 180 days prior to completion of second sputum collection for Xpert testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected pulmonary TB patients in Huashan Hospital, Wenzhou Central Hospital and Hangzhou Red Cross Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of clinically diagnosed TB participants with CRISPR-based test MTB positive in sputum/BALF who are Xpert MTB/RIF Assay positive and/or MGIT culture positive for M.tuberculosis. | week 0
Proportion of clinically diagnosed TB participants with CRISPR-based test MTB positive in sputum/BALF who are Xpert MTB/RIF Assay negative and/or MGIT culture negative for M.tuberculosis. | week 0
Proportion of clinically diagnosed non-TB participants with CRISPR-based test MTB positive in sputum/BALF. | week 0

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zifodya JS, Kreniske JS, Schiller I, Kohli M, Dendukuri N, Schumacher SG, Ochodo EA, Haraka F, Zwerling AA, Pai M, Steingart KR, Horne DJ. Xpert Ultra versus Xpert MTB/RIF for pulmonary tuberculosis and rifampicin resistance in adults with presumptive pulmonary tuberculosis. Cochrane Database Syst Rev. 2021 Feb 22;2(2):CD009593. doi: 10.1002/14651858.CD009593.pub5. PMID 33616229